CLINICAL TRIAL: NCT04672239
Title: A Proof-of-concept RCT of Version 3.0 of the Smoking Cessation Smartphone App "Smiling Instead of Smoking" (SiS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Bettina B. Hoeppner, Associate Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020P003466
Record Dates: First submitted 2020-12-10; First posted 2020-12-17 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Nondaily Smoking
Keywords: nondaily smoking; smartphone app; smoking cessation; QuitGuide; Smiling instead of Smoking; SiS; positive psychology; mHealth
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: 3-group proof-of-concept RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Smiling Instead of Smoking (SiS) app (Experimental): Participants will be onboarded (remotely) to the smartphone app "Smiling instead of Smoking" (SiS), and will be asked to use it for 7 weeks while they quit smoking.
  Interventions: Behavioral: Smartphone app "Smiling instead of Smoking" (SiS) Version 3
- QuitGuide (QG) app (Active Comparator): Participants will be onboarded (remotely) to the smartphone app "QuitGuide" (QG), and will be asked to use it for 7 weeks while they quit smoking.
  Interventions: Behavioral: Smartphone app "QuitGuide" (QG)
- Clearing the Air (CTA) brochure (Other): Participants will be onboarded (remotely) to the NCI brochure "Clearing the Air" (CTA), and will be asked to use it for 7 weeks while they quit smoking.
  Interventions: Behavioral: Brochure "Clearing the Air" (CTA)

INTERVENTIONS:
Behavioral: Smartphone app "Smiling instead of Smoking" (SiS) Version 3 — Participants will be onboarded to the smartphone app SiS and will be asked to use it for 7 weeks to support them in quitting smoking.
  Other Names: SiS
  Arms: Smiling Instead of Smoking (SiS) app
Behavioral: Smartphone app "QuitGuide" (QG) — Participants will be onboarded to the NCI smartphone app QG and will be asked to use it for 7 weeks to support them in quitting smoking.
  Other Names: QG
  Arms: QuitGuide (QG) app
Behavioral: Brochure "Clearing the Air" (CTA) — Participants will be onboarded to the brochure "Clearing the Air" and will be asked to use it for 7 weeks to support them in quitting smoking.
  Arms: Clearing the Air (CTA) brochure

SUMMARY:
This is the third study in a series of 3 studies to develop a smartphone app to support nondaily smokers in quitting smoking, as funded by the American Cancer Society grant #RSG CPPB - 130323 (project dates: 07/01/2017 - 6/30/2021). Study 1 (2017P001106) demonstrated feasibility and acceptability when smokers were onboarded in person. Study 2 (2018P002699) demonstrated feasibility and acceptability when smokers were onboarded remotely, nationwide. The present study is Study 3. It is a 3-group proof-of-concept RCT, in which we seek to test if our app (i.e., Version 3 of our developed smartphone app, called 'Smiling instead of Smoking' (SiS)) is superior to treatment as usual (i.e., TAU) and superior to a control app (i.e., the National Cancer Institute's smartphone app "QuitGuide" (QG).

DETAILED DESCRIPTION:
This is a nation-wide proof-of-concept randomized controlled trial conducted entirely remotely. Participation will last 6 months and entails:

* Completing a scripted onboarding call (approximately 30-45 minutes)
* Making a quit attempt
* Engaging with smoking cessation support (randomized) over the course of seven weeks, one week prior and 6 weeks following the originally chosen quit day
* Completing five online, REDCap-administered surveys, administered prior to the quit day (online, as part of a screening test), and at 2-week, 6-week, 3-month, and 6-month follow-ups of the participant's chosen quit day

The Aims of the study are:

1. Test for differences between randomized groups on the primary outcome (i.e., self-efficacy to remain abstinent, as measured via the Smoking Self-Efficacy Questionnaire), as measured at end of treatment (i.e., 6 weeks after the participants' chosen smoking quit day)
2. Test for differences between randomized groups on secondary outcomes (as listed in Detailed Protocol)
3. (exploratory) To test, via mediational modeling, how treatment via the proposed app conferred benefit; or, if not effective, if failure is due to the treatment failing to impact hypothesized mechanisms of change, or because these mechanisms fail to impact outcome.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years of age
* smartphone ownership (Android or iPhone only)
* current nondaily smoker, who smokes at least weekly, and no more than 25 out of the past 30 days
* lifetime history of having smoked 100+ cigarettes
* willing to make a smoking quit attempt
* currently residing in the United States of America

Exclusion Criteria:

* Under 18 years of age
* Does not own an Android or iPhone
* Is not a nondaily smoker, who smokes at least weekly, and no more than 25 out of the past 30 days
* Does not have a lifetime history of having smoked 100+ cigarettes
* Is not willing to make a smoking quit attempt
* Is not currently residing in the United States of America

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2021-01-28 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2023-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Hoeppner, Ph.D., M.S., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share IPD

REFERENCES:
- [Background] Etter JF, Bergman MM, Humair JP, Perneger TV. Development and validation of a scale measuring self-efficacy of current and former smokers. Addiction. 2000 Jun;95(6):901-13. doi: 10.1046/j.1360-0443.2000.9569017.x. PMID 10946439
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Adler MG, Fagley NS. Appreciation: individual differences in finding value and meaning as a unique predictor of subjective well-being. J Pers. 2005 Feb;73(1):79-114. doi: 10.1111/j.1467-6494.2004.00305.x. PMID 15660674
- [Background] Brooke J. SUS-A quick and dirty usability scale. Usability evaluation in industry. 1996;189(194):4-7.
- [Derived] Hoeppner BB, Siegel KR, Futter AE, Finley-Abboud D, Williamson AC, Kahler CW, Park ER, Hoeppner SS. Smoking Cessation Smartphone App for Nondaily Smoking With Telephone Onboarding: Proof-of-Concept Randomized Controlled Trial. JMIR Mhealth Uhealth. 2025 Jan 15;13:e53971. doi: 10.2196/53971. PMID 39814363
- [Derived] Hoeppner BB, Siegel KR, Dickerman SR, Todi AA, Kahler CW, Park ER, Hoeppner SS. Testing the Outcomes of a Smoking Cessation Smartphone App for Nondaily Smokers: Protocol for a Proof-of-concept Randomized Controlled Trial. JMIR Res Protoc. 2023 Feb 14;12:e40867. doi: 10.2196/40867. PMID 36787172

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant in each treatment arm decided against the study during the onboarding process and before starting any study procedures. These were excluded from analysis in a modified intent to treat approach for an enrolled and active sample of n=226.
Groups:
- SiS App Treatment: Participants were onboarded (remotely) to the smartphone app "Smiling instead of Smoking" (SiS) Version 3, and were asked to use it for 7 weeks while they quit smoking.
- QG App Treatment: Participants were onboarded (remotely) to the National Cancer Institute's (NCI) smartphone app "QuitGuide" (QG), and were asked to use it for 7 weeks while they quit smoking.
- CTA Pamphlet: Participants were onboarded (remotely) to the National Cancer Institute's (NCI) brochure "Clearing the Air" (CTA), and were asked to use it for 7 weeks while they quit smoking.
Period: Week 2 Survey
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Started | 80 | 75 | 71
Completed | 69 | 69 | 59
Not Completed | 11 | 6 | 12
Not completed — Failed survey check items | 1 | 2 | 3
Not completed — Partially completed survey | 7 | 1 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 2 | 5
Period: Week 6 Survey
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Started (All participants who did not withdraw themselves or were not withdrawn by the PI were automatically invited to complete any follow-up survey, even if they missed, failed a check-item on, or only partially completed a previous survey.) | 80 | 74 (Cumulatively, 1 participant had withdrawn prior to the week 6 survey.) | 71
Completed | 62 | 65 | 61
Not Completed | 18 | 9 | 10
Not completed — Failed survey check items | 2 | 2 | 2
Not completed — Partially completed survey | 3 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Withdrawn by PI | 0 | 1 | 0
Not completed — Lost to Follow-up | 12 | 2 | 5
Period: 3-Month Follow-up Survey
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Started (All participants who did not withdraw themselves or were not withdrawn by the PI were automatically invited to complete any follow-up survey, even if they missed, failed a check-item on, or only partially completed a previous survey.) | 79 (Cumulatively, 1 participant had withdrawn prior to the 3-month follow-up survey.) | 72 (Cumulatively, 3 participants had withdrawn themselves or were withdrawn by the PI prior to the 3-month follow-up survey.) | 70 (Cumulatively, 1 participant had withdrawn prior to the 3-month follow-up survey.)
Completed | 57 | 62 | 53
Not Completed | 22 | 10 | 17
Not completed — Failed survey check items | 2 | 3 | 2
Not completed — Partially completed survey | 3 | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 1
Not completed — Lost to Follow-up | 17 | 5 | 11
Period: 6-Month Follow-up Survey
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Started (All participants who did not withdraw themselves or were not withdrawn by the PI were automatically invited to complete any follow-up survey, even if they missed, failed a check-item on, or only partially completed a previous survey.) | 79 (Cumulatively, 1 participant had withdrawn prior to the 6-month follow-up survey.) | 71 (Cumulatively, 4 participants had withdrawn or were withdrawn prior to the 6-month follow-up survey.) | 69 (Cumulatively, 2 participants had withdrawn prior to the 6-month follow-up survey.)
Completed | 57 | 59 | 58
Not Completed | 22 | 12 | 11
Not completed — Failed survey check items | 2 | 0 | 0
Not completed — Partially completed survey | 7 | 0 | 2
Not completed — Lost to Follow-up | 13 | 12 | 9

BASELINE CHARACTERISTICS:
Population: All randomized and starting study procedures (n=226; see Participant flow pre-assignment details). Some measures had missing data.
Groups:
- Total: Total of all reporting groups
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet | Total
Number analyzed (Participants) | 80 | 75 | 71 | 226
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.1) | 41.6 (13.1) | 40.0 (12.5) | 41.0 (12.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 28 | 37 | 30 | 95
  Female | 51 | 36 | 41 | 128
  Other | 1 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 16 | 6 | 37
  Not Hispanic or Latino | 62 | 57 | 64 | 183
  Unknown or Not Reported | 3 | 2 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 23 | 19 | 13 | 55
  White | 50 | 46 | 48 | 144
  More than one race | 4 | 6 | 4 | 14
  Unknown or Not Reported | 2 | 3 | 1 | 6
Highest level of education completed [Count of Participants; unit: Participants] — Data was collected via self-report in pre-specified categories.
  Participants
    High School or less | 7 | 12 | 15 | 34
    Some college | 31 | 38 | 25 | 94
    College degree or higher | 42 | 25 | 30 | 97
    Declined to answer | 0 | 0 | 1 | 1
Employment [Count of Participants; unit: Participants] — Collected via self-report with pre-specified categories.
  Participants
    Full-time | 29 | 30 | 27 | 86
    Part-time | 14 | 11 | 18 | 43
    Unemployed | 32 | 33 | 23 | 88
    Declined to answer | 5 | 1 | 3 | 9
Household Income [Count of Participants; unit: Participants] — Collected via self-report with pre-specified categories.
  Participants
    $39,999 or less | 41 | 42 | 30 | 113
    $40,000 - 69,999 | 18 | 18 | 22 | 58
    $70,000 - 99,999 | 16 | 8 | 10 | 34
    $100,000 or more | 4 | 7 | 8 | 19
    Declined to answer | 1 | 0 | 1 | 2
Rurality [Count of Participants; unit: Participants] — Collected via self-report with pre-specified categories.
  Participants
    Urban | 39 | 34 | 27 | 100
    Suburban | 29 | 24 | 35 | 88
    Rural | 12 | 17 | 9 | 38
US region [Count of Participants; unit: Participants] — Collected via self-report with pre-specified categories.
  Participants
    Northeast | 22 | 15 | 14 | 51
    Midwest | 10 | 11 | 10 | 31
    South | 34 | 34 | 29 | 97
    West | 14 | 15 | 18 | 47
Number of days smoked in past 30 days [Mean (Standard Deviation); unit: number of days] — Population: Some participants declined to answer this question.
  number of days
    number analyzed (Participants) | 77 | 75 | 71 | 223
    (all) | 15.3 (5.4) | 14.7 (4.8) | 14.6 (4.5) | 14.9 (4.9)
Cigarettes per smoking day [Mean (Standard Deviation); unit: cigarettes per day] — Population: Some participants declined to answer this question.
  cigarettes per day
    number analyzed (Participants) | 74 | 69 | 66 | 209
    (all) | 3.5 (2.9) | 3.0 (2.2) | 3.8 (3.0) | 3.4 (2.7)
Fagerstrom Test for Nicotine Dependence, total score [Median (Inter-Quartile Range); unit: units on a scale] — The Fagerström Test for Nicotine Dependence is a standard instrument for assessing the intensity of physical addiction to nicotine. The test contains six items that evaluate the quantity of cigarette consumption, the compulsion to use, and dependence.
  In scoring the Fagerstrom Test for Nicotine Dependence, yes/no items are scored from 0 to 1 and multiple-choice items are scored from 0 to 3. The items are summed to yield a total score of 0-10. The higher the total Fagerström score, the more intense is the patient's physical dependence on nicotine. Population: One participant missed one or more items on the scale.
  units on a scale
    number analyzed (Participants) | 79 | 75 | 71 | 225
    (all) | 1.0 [0.0 to 4.0] | 1.0 [0.0 to 3.0] | 1.0 [0.0 to 3.0] | 1.0 [0.0 to 3.0]
Ever smoked daily? [Count of Participants; unit: Participants]
  Yes | 54 | 53 | 44 | 151
  No | 25 | 22 | 27 | 74
  Declined to answer | 1 | 0 | 0 | 1
Ever tried to quit smoking before [Count of Participants; unit: Participants] — Collected via self-report with pre-specified categories.
  Participants
    Yes | 49 | 56 | 52 | 157
    No | 31 | 19 | 19 | 69
Ever used electronic cigarettes [Count of Participants; unit: Participants] — Collected via self-report with pre-specified categories.
  Participants
    Yes | 46 | 41 | 46 | 133
    No | 34 | 34 | 25 | 93
Currently uses electronic cigarettes [Count of Participants; unit: Participants]
  Yes | 14 | 10 | 9 | 33
  No | 66 | 65 | 62 | 193
CES-D total scores [Median (Inter-Quartile Range); unit: units on a scale] — The Center for Epidemiologic Studies Depression Scale (CES-D) is a 20-item scale with Likert scales ranging from "rarely or none of the time (less than 1 day)" to "Most or all of the time (5-7 days)". The possible range of scores is zero to 60, with higher scores indicating greater depression severity.
  units on a scale | 8.0 [4.5 to 12.5] | 9.0 [5.0 to 16.0] | 11.0 [6.0 to 15.0] | 9.0 [5.0 to 15.0]
GAD-7 total scores [Mean (Standard Deviation); unit: units on a scale] — The Generalized Anxiety Disorder 7-item (GAD-7) scale is a easy to perform initial screening tool for generalized anxiety disorder. Items are score on 4-point Likert scales ranging from "Not at all" to "Nearly every day". GAD-7 total scores range from 0 to 21, with higher values indicating greater depression severity.
  units on a scale | 5.7 (4.8) | 6.5 (5.4) | 7.2 (5.1) | 6.4 (5.1)
GSES total scores [Mean (Standard Deviation); unit: units on a scale] — The General Self-Efficacy Scale (GSES) is a 10 item scale that is rated on 4-point Likert scales ranging from "Not at all true" to "Exactly true". Total scores range from 10 to 40, with higher scores indicating greater general self-efficacy.
  units on a scale | 31.9 (5.0) | 31.7 (4.9) | 30.8 (4.7) | 31.5 (4.9)
Anhedonia [Count of Participants; unit: Participants] — The Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item scale for the assessment of hedonic tone. Each item has four possible responses: strongly disagree, disagree, agree, or strongly agree. Either of the "disagree" responses score one point, and either of the "agree" responses score 0 points. Total scores can range from 0 to 14 with higher scores indicating greater anhedonia (i.e., smaller capacity to experience pleasure). Scores were recoded to indicate to indicate whether people had possible indication of anhedonia (scores > 2) or not. Population: Two participants (1 from SiS App Treatment, 1 from CTA Pamphlet) missed two or more items on the scale, and scale scores were not calculated for them.
  Participants
    Yes: number analyzed (Participants) | 79 | 75 | 70 | 224
    Yes | 11 | 18 | 17 | 46
    No: number analyzed (Participants) | 79 | 75 | 70 | 224
    No | 68 | 57 | 53 | 178
Ever told they had a mental health or psychological condition [Count of Participants; unit: Participants] — Asked as a Yes/No question.
  Participants
    Yes | 24 | 23 | 22 | 69
    No | 56 | 52 | 49 | 157
SIMP - Extraversion [Mean (Standard Deviation); unit: units on a scale] — Extraversion was measured on a Single-Item Measures of Personality (SIMP) scale measured on 9-point Likert scale that ranged from "someone who is a reserved, private person, doesn't like to draw attention to themselves and can be shy around strangers" (=1) to "someone who is talkative, outgoing, is comfortable around people, but could be noisy and attention seeking" (=9)
  units on a scale | 5.5 (2.1) | 5.2 (2.5) | 5.1 (2.5) | 5.3 (2.4)
SIMP - Agreeableness [Mean (Standard Deviation); unit: units on a scale] — Agreeableness was measured on a Single-Item Measures of Personality (SIMP) scale measured on 9-point Likert scale that ranged from "someone who is forthright, tends to be critical and find fault with others and doesn't suffer fools gladly" (=1) to "someone who is generally trusting and forgiving, is interested in people, but can be taken for granted and finds it difficult to say no" (=9)
  units on a scale | 6.6 (1.9) | 6.2 (2.4) | 6.4 (2.1) | 6.4 (2.1)
SIMP - Emotional stability [Mean (Standard Deviation); unit: units on a scale] — Emotional stability was measured on a Single-Item Measures of Personality (SIMP) scale measured on 9-point Likert scale that ranged from "someone who is sensitive and excitable, and can be tense" (=1) to "someone who is relaxed, unemotional, rarely gets irritated and seldom feels blue" (=9)
  units on a scale | 5.1 (2.4) | 4.7 (2.2) | 4.4 (1.9) | 4.8 (2.2)
SIMP - Conscientiousness [Mean (Standard Deviation); unit: units on a scale] — Conscientisousness was measured on a Single-Item Measures of Personality (SIMP) scale measured on 9-point Likert scale that ranged from "someone who doesn't necessarily work on a schedule, tends to be flexible, but disorganised and often forgets to put things back in their proper place" (=1) to "someone who likes to plan things, likes to tidy up, pays attention to details, but can be rigid or inflexible" (=9)
  units on a scale | 5.2 (2.6) | 5.2 (2.3) | 5.7 (2.3) | 5.4 (2.4)
SIMP - Openness [Mean (Standard Deviation); unit: units on a scale] — Openness was measured on a Single-Item Measures of Personality (SIMP) scale measured on 9-point Likert scale that ranged from "someone who spends time reflecting on things, has an active imagination and likes to think of new ways of doing things, but may lack pragmatism" (=1) to "someone who is a practical person who is not interested in abstract ideas, prefers work that is routine and has few artistic interests" (=9)
  units on a scale | 3.9 (2.1) | 3.6 (2.0) | 4.1 (2.3) | 3.9 (2.1)
Any alcohol in the past 30 days [Count of Participants; unit: Participants] — Asked as a Yes/No question
  Participants
    Yes | 45 | 37 | 40 | 122
    No | 35 | 38 | 31 | 104
Any weeks of exceeding the drinking guidelines in the past 30 days [Count of Participants; unit: Participants] — Using part of the the National Institute on Alcohol Abuse and Alcoholism (NIAAA) guidelines:
  For men, consuming more than 14 drinks per week For women, consuming more than 7 drinks per week
  Participants
    Yes | 23 | 18 | 19 | 60
    No | 57 | 57 | 52 | 166
Any binge drinking in the past 30 days [Count of Participants; unit: Participants] — Using the definition of the Substance Abuse and Mental Health Services Administration (SAMHSA), which conducts the annual National Survey on Drug Use and Health (NSDUH), which defines binge drinking as 5 or more alcoholic drinks for males or 4 or more alcoholic drinks for females on the same occasion (i.e., at the same time or within a couple of hours of each other) on at least 1 day in the past month.
  Participants
    Yes | 25 | 15 | 18 | 58
    No | 55 | 60 | 53 | 168

OUTCOME MEASURES:

1. Primary Outcome: End of Treatment Group Differences in Smoking Self-Efficacy Questionnaire (SEQ)
Description: The Smoking Self-Efficacy Questionnaire (SEQ-12) (Etter, Bergman, Humair, & Perneger, 2000) is a two-dimensional 12-item self-report scale measuring a person's confidence in his or her ability to abstain from smoking when facing internal stimuli (e.g. feeling depressed) and external stimuli (e.g. being with smokers) on a 0-100 slider scale (i.e., 0=not at all confident that I can refrain; 100=extremely confident that I can refrain). Scale scores are created by mean scoring across items and range from 0 to 100. Higher scores indicate greater self-efficacy to abstain from smoking.
Time Frame: Up to 24 weeks post quit day. Note that the 7 weeks of treatment started 1 week prior to the quit date (baseline = week -1).
Population: Some participants had missing data at various assessment time-points, but all enrolled participants provided data for at least one assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Smiling Instead of Smoking: Participants will be onboarded (remotely) to the smartphone app "Smiling instead of Smoking" (SiS), and will be asked to use it for 7 weeks while they quit smoking.
  Smartphone app "Smiling instead of Smoking" (SiS) Version 3: Participants will be onboarded to the smartphone app SiS and will be asked to use it for 7 weeks to support them in quitting smoking.
- Quit Guide: Participants will be onboarded (remotely) to the smartphone app "QuitGuide" (QG), and will be asked to use it for 7 weeks while they quit smoking.
  Smartphone app "QuitGuide" (QG): Participants will be onboarded to the NCI smartphone app QG and will be asked to use it for 7 weeks to support them in quitting smoking.
- Clearing the Air: Participants will be onboarded (remotely) to the NCI brochure "Clearing the Air" (CTA), and will be asked to use it for 7 weeks while they quit smoking.
  Brochure "Clearing the Air" (CTA): Participants will be onboarded to the brochure "Clearing the Air" and will be asked to use it for 7 weeks to support them in quitting smoking.
Arm/Group | Smiling Instead of Smoking | Quit Guide | Clearing the Air
Number analyzed (Participants) | 80 | 75 | 71
units on a scale
  Baseline: number analyzed (Participants) | 78 | 72 | 69
  Baseline | 63.81 (17.24) | 60.74 (16.67) | 58.45 (19.10)
  Week 2 post-quit: number analyzed (Participants) | 74 | 68 | 55
  Week 2 post-quit | 71.79 (18.56) | 67.58 (15.69) | 65.40 (16.59)
  Week 6 post-quit: number analyzed (Participants) | 64 | 66 | 61
  Week 6 post-quit | 78.34 (17.31) | 71.34 (17.67) | 68.99 (19.80)
  Week 12 post-quit (3-month follow-up): number analyzed (Participants) | 60 | 63 | 56
  Week 12 post-quit (3-month follow-up) | 81.16 (17.35) | 76.20 (19.50) | 75.22 (19.12)
  Week 24 post-quit (6-month follow-up): number analyzed (Participants) | 61 | 59 | 60
  Week 24 post-quit (6-month follow-up) | 80.23 (18.41) | 80.51 (20.33) | 74.48 (23.42)
Statistical Analysis 1: Comparison: Smiling Instead of Smoking vs Quit Guide; This proof-of-concept RCT was powered to detect an effect size of d=0.50 between SiS3 and either of the two control groups. Using SAS PROC POWER, it was determined that a sample size of n=64 per group would be needed to detect this effect in a 2-sided t-test with p=.05. Assuming a retention rate of 85%, it was determined that one needed to enroll n=75 per group in order to retain n=64 by end of treatment; Test type: Superiority; p = 0.0219, Mixed Models Analysis — We used hierarchical linear mixed models with maximum likelihood estimation of all available longitudinal data to handle missing data, then used a planned, pairwise comparison to test for end-of-treatment group differences; Mean Difference (Final Values) = 7.3341, 95% CI 2-sided [1.0734 to 13.5948] — Model-estimated difference for the pairwise group difference at week 6 post-quit (end-of-treatment)
Statistical Analysis 2: Comparison: Smiling Instead of Smoking vs Clearing the Air; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0072, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 8.7775, 95% CI 2-sided [2.4070 to 15.1480] — Model-estimated difference for the pairwise group difference at week 6 post-quit (end-of-treatment)

2. Secondary Outcome: Self-reported 30-day Point-prevalence Abstinence
Description: Participants responded to the multiple choice question, "What is your current smoking status?" with answer options: "I smoke daily", "I smoke non-daily (and have smoked in the past 7 days)", "I smoke nondaily (but have NOT smoked in the past 7 days)", and "I do not smoke at all"). If participants reported that they did not smoke at all, they were asked: "Have you been abstinent during the past 30 days?" (yes/no). All participants who reported smoking daily or nondaily to the first question, or who reported not smoking at all but had smoking in the past 30 days, or those who left either of those questions unanswered were marked as NOT 30-day point prevalent smoking abstinent (not included in the abstinent count below). People who reported not smoking at all and being smoking-abstinent for the past 30 days were marked as 30-day point prevalent smoking abstinent (include in the abstinent count below).
Time Frame: Assessed at 2, 6, 12, and 24 weeks post-quit day. Note that the 7 weeks of treatment started 1 week prior to the quit date (i.e., baseline = week -1).
Population: Participants with missing data were assumed to be smoking (i.e., not 30-day point-prevalent abstinent from smoking).
Measure: Count of Participants; unit: Participants
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Number analyzed (Participants) | 80 | 75 | 71
Participants
  Week 2 post-quit | 9 | 3 | 9
  Week 6 post-quit | 32 | 23 | 18
  Week 12 post-quit (3-month follow-up) | 36 | 31 | 21
  Week 24 post-quit (6-month follow-up) | 38 | 32 | 31
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; This was an exploratory aim, so no power analysis was conducted. We hypothesized, that the 30-day point prevalence smoking cessation prevalence would be higher in the SiS app treatment compared to the QuitGuide app treatment. Participants with missing data were assumed to be smoking. We modeled all available data over time and present the cross-sectional group difference test at week 6 post quit (i.e., end-of-treatment); Test type: Superiority; p = 0.2259, Generalized Linear Model; We used a Generalized Linear Model with binomial distribution (abstinent vs. smoking) and logit link with repeated measures over time; Odds Ratio (OR) = 1.5072, 95% CI 2-sided [0.7759 to 2.9281] — The odds ratio compares the SiS app treatment to the QG app treatment at week 6 post-quit (end-of-treatment)
Statistical Analysis 2: Comparison: SiS App Treatment vs CTA Pamphlet; This was an exploratory aim, so no power analysis was conducted. We hypothesized, that the 30-day point prevalence smoking cessation prevalence would be higher in the SiS app treatment compared to the Clearing the Air pamphlet treatment. Participants with missing data were assumed to be smoking. We modeled all available data over time and present the cross-sectional group difference test at week 6 post quit (i.e., post-treatment); Test type: Superiority; p = 0.0579, Generalized Linear Model; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 1.9630, 95% CI 2-sided [0.9776 to 3.9415] — The odds ratio compares the SiS app treatment to the CtA pamphlet at week 6 post-quit (end-of-treatment)

3. Secondary Outcome: Self-reported Past Week Cigarette Change
Description: If participants report having smoked in the past 7 days, they were asked to indicate how many cigarettes they smoked each day ("Last Monday:, Last Sunday:). Changes in cigarette consumption were calculated by subtracting the number of cigarettes smoked in the week leading up to the baseline assessment, as measured in the baseline survey, from the number of cigarettes smoked in the week leading up to the 2, 6, 12, and 24 week post-quit assessments, as assessed in these respective surveys.
Time Frame: as for outcome 2
Population: All available survey data at each assessment was used; by week 2 post-quit several participants had missing data for that and all subsequent assessments (n=3 for the SiS app, n=2 for the QG app, and n=3 for the CTA pamphlet groups).
Measure: Median (Inter-Quartile Range); unit: Change in weekly cigs since baseline
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Number analyzed (Participants) | 77 | 73 | 68
Change in weekly cigs since baseline
  Week 2 post-quit: number analyzed (Participants) | 76 | 70 | 63
  Week 2 post-quit | -6.0 [-12.0 to -2.5] | -6.0 [-11.0 to -3.0] | -7.0 [-11.0 to -3.0]
  Week 6 post-quit: number analyzed (Participants) | 65 | 67 | 63
  Week 6 post-quit | -5.0 [-12.0 to -1.0] | -6.0 [-11.0 to -3.0] | -7.0 [-13.0 to -4.0]
  Week 12 post-quit (3-month follow-up): number analyzed (Participants) | 60 | 63 | 56
  Week 12 post-quit (3-month follow-up) | -6.0 [-12.0 to -1.5] | -6.0 [-11.0 to -2.0] | -7.0 [-13.5 to -3.0]
  Week 24 post-quit (6-month follow-up): number analyzed (Participants) | 63 | 59 | 60
  Week 24 post-quit (6-month follow-up) | -6.0 [-9.5 to 0.0] | -6.0 [-10.0 to -2.0] | -7.0 [-12.5 to -2.0]
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.9152, Wilcoxon (Mann-Whitney); Pairwise Two-Sided Multiple Comparison Analysis Dwass, Steel, Critchlow-Fligner Method; Wilcoxon Z = 0.4010 — SiS app treatment vs. QuitGuide app treatment at week 6 post-quit (end-of-treatment)
Statistical Analysis 2: Comparison: SiS App Treatment vs CTA Pamphlet; Test type: Superiority; p = 0.3557, Wilcoxon (Mann-Whitney); Pairwise Two-Sided Multiple Comparison Analysis Dwass, Steel, Critchlow-Fligner Method; Wilcoxon Z = 1.3720 — Pairwise comparison, SiS app treatment vs. CTA pamphlet at week 6 post-quit (end-of-treatment)

4. Secondary Outcome: Satisfaction With Smoking Cessation Support
Description: As measured using the Client Satisfaction Scale (CSQ-8) (Larsen, 1979), an 8 item multiple choice measure that will be used to assess participants' satisfaction with the smoking cessation support they receive (e.g., "How satisfied are you with the amount of help you received?"). Scores are summed across items and range from 8 to 32, with higher scores indicating greater satisfaction.
Time Frame: Assessed at treatment end (week 6 post-quit). Note that the 7 weeks of treatment started 1 week prior to the quit date (i.e., baseline = week -1).
Population: Participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Clearing the Air Pamphlet: Participants were onboarded (remotely) to the National Cancer Institute's (NCI) brochure "Clearing the Air" (CTA), and were asked to use it for 7 weeks while they quit smoking.
Arm/Group | SiS App Treatment | QG App Treatment | Clearing the Air Pamphlet
Number analyzed (Participants) | 65 | 67 | 63
units on a scale | 26.91 (5.30) | 26.61 (4.51) | 25.65 (5.80)
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.7469, t-test, 2 sided — The p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.2936, 95% CI 2-sided [-1.4983 to 2.0856] — Comparison of SiS app treatment to the QuitGuide treatment as control (Contrast coding SiS 1, QG -1)
Statistical Analysis 2: Comparison: SiS App Treatment vs Clearing the Air Pamphlet; Test type: Superiority; p = 0.1747, t-test, 2 sided — The p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 1.2569, 95% CI 2-sided [-0.5628 to 3.0766] — Comparison of SiS app treatment to the Clearing the Air pamphlet treatment as control (Contrast coding SiS 1, CtA -1)

5. Secondary Outcome: Time Spent Applying Content Brought up by the Apps/"Clearing the Air"
Description: Measured using the following single item, "During this past week, how much time did you spend applying or contemplating the content of the SiS app/QG app/"Clearing the Air"?" [in minutes].
Time Frame: as for outcome 4
Population: Participants with missing data were excluded from analysis.
Measure: Median (Inter-Quartile Range); unit: minutes per week
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Number analyzed (Participants) | 64 | 66 | 63
minutes per week | 30.0 [29.0 to 70.0] | 25.0 [10.0 to 60.0] | 30.0 [10.0 to 60.0]
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.1315, Wilcoxon (Mann-Whitney) — p-values were not adjusted for multiple comparisons; Pairwise Two-Sided Multiple Comparison Analysis Dwass, Steel, Critchlow-Fligner Method; Wilcoxon Z = 1.9255
Statistical Analysis 2: Comparison: SiS App Treatment vs CTA Pamphlet; Test type: Superiority; p = 0.3403, Wilcoxon (Mann-Whitney) — the p-value was not adjusted for multiple comparisons; Pairwise Two-Sided Multiple Comparison Analysis Dwass, Steel, Critchlow-Fligner Method; Wilcoxon Z = 1.4010 — SiS app vs. Clearing the Air pamphlet

6. Secondary Outcome: Use of Smoking Cessation Strategies
Description: Assessed using a study-specific, unpublished 8-item measure in which participants rated the extent to which they agreed or disagreed with statements about the smoking cessation support they received and the things they did while quitting (5-point Likert scale, 1=strongly disagree, 5=strongly agree, e.g., "I used [the assigned treatment] the way I was supposed to (in the days leading up to and following my quit attempt)." and "I avoided situations that would make me want to smoke."). The scores of the 8 items were averaged, so that scores could range from 1 to 5, where higher scores indicate stronger agreement with the use of a larger combination of smoking cessation strategies (i.e., a more positive outcome).
Time Frame: as for outcome 4
Population: Participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Number analyzed (Participants) | 63 | 65 | 61
units on a scale | 4.13 (0.63) | 3.90 (0.59) | 3.97 (0.69)
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.0429, t-test, 2 sided — p-value is not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.2289, 95% CI 2-sided [0.007364 to 0.4505]; SiS app vs. QuitGuide app
Statistical Analysis 2: Comparison: SiS App Treatment vs CTA Pamphlet; Test type: Superiority; p = 0.1600, t-test, 2 sided — p-value is not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.1609, 95% CI 2-sided [-0.06415 to 0.3860]; SiS app vs. CtA pamphlet

7. Secondary Outcome: Perceived Impact of the Provided Materials on Quitting
Description: Assessed using a study-specific, unpublished 17-item measure in which participants rated the extent to which they agreed or disagreed with statements about the helpfulness of their assigned app during the quitting process (e.g., "[the app]...gave me confidence that I can quit smoking.", "[the app]... made me feel that I knew the right steps to take to quit.", and "[the app] ...reminded me in crucial moments to stay quit."). Items were rated on 5-point Likert scales ranging from 1="strongly disagree" to 5="strongly agree". The scores of the 17 items were averaged, so that scores could range from 1 to 5, where higher scores indicate stronger agreement with perceived impact of the smoking cessation support their assigned app provided (i.e., a more positive outcome).
Time Frame: as for outcome 4
Population: Participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 4.13 (0.72) | 3.98 (0.55) | 3.84 (0.73)
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.1996, t-test, 2 sided — p-value is not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.1520, 95% CI 2-sided [-0.08092 to 0.3848]; SiS app vs. QG app
Statistical Analysis 2: Comparison: SiS App Treatment vs CTA Pamphlet; Test type: Superiority; p = 0.0154, t-test, 2 sided — p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 0.2920, 95% CI 2-sided [0.05636 to 0.5276]; SiS app vs. CtA pamphlet (control)

8. Secondary Outcome: Appreciation
Description: As measured using the Appreciation Scale, (Adler & Fagley, 2005) an 18-item scale assessing the degree to which one is appreciative. Ten of the items assess frequency of action (e.g., "I do things to remind myself to be thankful", using a 7-point Likert scale of: 1 = "More than once a day" to 7 = "Never"). The remaining eight items assess level of agreement with appreciative statements (e.g., "I feel that it is a miracle to be alive", using a 7-point Likert scale of: 1 = "Strongly agree" to 7 = "Strongly disagree"). Item scores were summed to a total score with a possible range from 18 to 126 where higher scores indicate greater appreciation.
Time Frame: as for outcome 4
Population: Participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SiS App Treatment | QG App Treatment | CTA Pamphlet
Number analyzed (Participants) | 64 | 66 | 63
units on a scale | 108.91 (13.46) | 106.28 (15.29) | 104.98 (14.26)
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.2988, t-test, 2 sided — p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 2.6255, 95% CI 2-sided [-2.3458 to 7.5968]; SiS app vs. QuitGuide app (control)
Statistical Analysis 2: Comparison: SiS App Treatment vs CTA Pamphlet; Test type: Superiority; p = 0.1251, t-test, 2 sided — p-value was not adjusted for multiple comparisons; Mean Difference (Final Values) = 3.9277, 95% CI 2-sided [-1.1015 to 8.9569]; SiS app vs. CtA pamphlet (control)

9. Secondary Outcome: Actual App Usage (SiS and QG Only)
Description: Number of days participants used the assigned app during the prescribed period of app use (i.e., 7 weeks for both apps). App usage is passively recorded by the app, which time-stamps every interaction with the app.
Time Frame: Cumulative from week 0 to week 24 post-quit day. Note that the 7 weeks of treatment started 1 week prior to the quit date (i.e., baseline = week -1).
Population: All participants randomized to either of the app treatment groups (SiS or QG).
Measure: Median (Inter-Quartile Range); unit: number of days of app use
Arm/Group | SiS App Treatment | QG App Treatment
Number analyzed (Participants) | 80 | 75
number of days of app use | 32.5 [11.0 to 39.5] | 26.0 [11.0 to 38.0]
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.4182, Wilcoxon (Mann-Whitney); Wilcoxon Z = -0.8096

10. Secondary Outcome: Self-reported App Usage, Weeks 3 to 6 Post-quit (SiS and QG Only)
Description: This was assessed via self-reported estimates of app use. Participants were asked on how many days they used the app in weeks 4, 5, and 6 post-quit ("On how many days per week did you use the app?"), and for how many minutes per typical day they used the assigned app ("On the days you used the app, how many minutes per day did you interact with the app?"). The days per week were multiplied by the minutes per app-use-day for each week, then averaged across the three weeks.
Time Frame: From week 3 to week 6 post-quit. Note that the 7 weeks of treatment started 1 week prior to the quit date (i.e., baseline = week -1).
Population: Participants with missing data were excluded.
Measure: Median (Inter-Quartile Range); unit: average minutes per week
Arm/Group | SiS App Treatment | QG App Treatment
Number analyzed (Participants) | 59 | 63
average minutes per week | 35.0 [21.0 to 70.0] | 22.5 [14.0 to 60.0]
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.0563, Wilcoxon (Mann-Whitney); Wilcoxon Z = 1.9090

11. Secondary Outcome: Likability Rating of the App (SiS and QG Only)
Description: Measured using the single item, "How much did you like using the smoking cessation app we asked you to use?" Participants respond on a 5-point Likert scale (1 = I strongly disliked using the app, 2 = I somewhat disliked using the app, 3 = I neither liked nor disliked using the app; 4 = I somewhat liked using the app, and 5 = I strongly liked using the app).
Time Frame: as for outcome 4
Population: Participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SiS App Treatment | QG App Treatment
Number analyzed (Participants) | 64 | 65
units on a scale | 4.19 (0.99) | 4.08 (0.87)
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.5018, t-test, 2 sided; Mean Difference (Final Values) = 0.1106, 95% CI 2-sided [-0.2143 to 0.4354]

12. Secondary Outcome: Satisfaction Rating of the Smoking Cessation Support (SiS and QG Only)
Description: Measured using the single item, "How satisfied are you with the smoking cessation support this app provided you with?" Participants respond on a 5-point Likert scale (1 = very unsatisfied, 2 = somewhat dissatisfied, 3 = neither satisfied nor dissatisfied, 4 = somewhat satisfied, 5 = very satisfied).
Time Frame: as for outcome 4
Population: Participants with missing data were excluded from analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SiS App Treatment | QG App Treatment
Number analyzed (Participants) | 64 | 64
units on a scale | 4.25 (1.04) | 4.11 (0.94)
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.4246, t-test, 2 sided; Mean Difference (Final Values) = 0.1406, 95% CI 2-sided [-0.2068 to 0.4880]

13. Secondary Outcome: App Usability Ratings (SiS and QG Only)
Description: As assessed via the System Usability Scale (SUS; Brooke, 1996), a ten-item attitude scale giving a global view of subjective assessments of usability, adapted to include language specific to the smoking app (e.g., "I found the smoking app unnecessarily complex" 5-point Likert: 1 = strongly disagree, 5 = strongly agree). Scale scores range from 0 to 100 with greater scores indicating a more favorable perception of usability of the app.
Time Frame: as for outcome 4
Population: Participants who were randomized to the two app treatment conditions (SiS and QuitGuide) and who completed the week 6 survey only.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SiS App Treatment | QG App Treatment
Number analyzed (Participants) | 63 | 65
units on a scale | 81.91 (17.10) | 79.48 (15.99)
Statistical Analysis 1: Comparison: SiS App Treatment vs QG App Treatment; Test type: Superiority; p = 0.4078, t-test, 2 sided; Mean Difference (Final Values) = 2.4296, 95% CI 2-sided [-3.3597 to 8.2188] — SiS app vs. QG (control)

ADVERSE EVENTS:
Time Frame: Adverse event data could be reported during the entire period of a participant's study participation (i.e., up to 6 months).
Description: Adverse events were not assessed systematically. However, they could be reported by spontaneous self-report by the participants at any point during the study.
Arm/Group | Smiling Instead of Smoking (SiS) App | QuitGuide (QG) App | Clearing the Air (CTA) Brochure
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/75 | 0/71
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/75 | 0/71
Other Adverse Events (participants affected / at risk) | 0/80 | 0/75 | 0/71

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT04672239/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT04672239/ICF_001.pdf